CLINICAL TRIAL: NCT04627402
Title: Effects of Adding Triamcinolone Acetonide to Conbercept in Diabetic Macular Edema With Limited Response to Anti-VEGF Treatment After One Injection
Brief Title: Effects of Adding Triamcinolone Acetonide to Conbercept Treatment for Refractory Diabetic Macular Edema (CONTE)
Acronym: CONTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Bingqian Liu, Associate Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020KYPJ127
Record Dates: First submitted 2020-10-29; First posted 2020-11-13 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2; Macular Edema
Keywords: diabetic macular edema; conbercept; triamcinolone acetonide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Macular Edema | interventions — KH902 fusion protein; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Diabetic macular edema.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection combo agents (Experimental): Intravitreous injection of triamcinolone acetonide (TA) and conbercept.
  Interventions: Drug: Conbercept and TA
- Injection single agent (Active Comparator): Intravitreous injection of conbercept only.
  Interventions: Drug: Conbercept

INTERVENTIONS:
Drug: Conbercept and TA — Intravitreous injection of Conbercept and TA
  Other Names: Combined agents
  Arms: Injection combo agents
Drug: Conbercept — Intravitreous injection of Conbercept
  Other Names: Single agent
  Arms: Injection single agent

SUMMARY:
This study aimed to compare intravitreous conbercept alone with conbercept plus intravitreous triamcinolone acetonide in DME eyes which showed limited response to anti-VEGF treatment after one injection.

DETAILED DESCRIPTION:
Some eyes with diabetic macular edema (DME) were not sensitive to anti-vascular endothelial growth factor (anti-VEGF) therapy and required continuous injections. Delayed control of macular edema might cause irreversible function loss. To predict the response to anti-VEGF treatment according to the CST change after one injection was proved reasonable recently. Adding intravitreous corticosteroids to the treatment regimen at early time might result in better outcomes than anti-VEGF therapy alone. Patients with diagnosis of refractory diabetic macular edema, confirmed by fluorangiography and optical coherence tomography (OCT), with limited response to one intravitreal anti-VEGF injection will be enrolled in the study. The enrolled patients will be randomized for the addition or not of the triamcinolone to intravitreal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes
* Vison decrease was mainly caused by diabetic macular edema (DME)
* BCVA of 20/800 to 20/40 (decimal)
* Central subfield retinal thickness (CST) ≥ 300μm by optical coherence tomography (OCT) in the study eye
* Pan-retinal photocoagulation finished at least 3 months ago, or no pan-retinal photocoagulation is expected in the next 6 months
* Within the last 3 months, one intravitreous injection of anti-VEGF agent was performed, the CST reduction one month after injection was ≤ 20%.

Exclusion Criteria:

* Non-DME related macular edema, or edema control would not benefit the vision (for example, macular atrophy)
* Exist of other reasons of macular edema, retinal vein occlusion, uveitis, iris rubeosis, high myopia
* Ocular media opacity of insufficient quality to obtain OCT images and fundus images in the study eye
* Intraocular or periorbital injection of steroids within the last 3 months
* Macular grid photocoagulation within the last 4 months
* History of vitrectomy
* History of scleral buckle within the last 4 months, or intraocular surgery is expected in the next 6 months
* Any sign of ocular infection, including conjunctivitis, hordeolum, dacryocystitis
* Myocardial infarction, heart failure, stroke, or transient ischemic attack within one month
* Pregnant or breastfeeding women
* Uncontrolled hypertension, or blood pressure >180/110
* Patients with uncontrolled hyperglycemia, or Hemoglobin A1C (HbA1c) ≥10.0%, or under hemodialysis , or started insulin usage within the last 4 months, or expected to start insulin use for hyperglycemia control in the next 4 months
* Those cannot follow visits on time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Macular thickness | 24 weeks
  Change in mean central subfield thickness from randomization visit measured with optical coherence tomography.

SECONDARY OUTCOMES:
Best-corrected visual acuity (BCVA) | 48 weeks
  Change in BCVA letter score from randomization visit as measured by the Early Treatment Diabetic Retinopathy Study (ETDRS).
Treatment number | 48 weeks
  The number of intravitreous injection treatments
Incidence of complications | 48 weeks
  The incidence of cataract and glaucoma

CONTACTS AND LOCATIONS:
Overall Officials: Bingqian Liu, MD, PhD, Principal Investigator — Zhongshan Ophthamic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Opthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maturi RK, Glassman AR, Liu D, Beck RW, Bhavsar AR, Bressler NM, Jampol LM, Melia M, Punjabi OS, Salehi-Had H, Sun JK; Diabetic Retinopathy Clinical Research Network. Effect of Adding Dexamethasone to Continued Ranibizumab Treatment in Patients With Persistent Diabetic Macular Edema: A DRCR Network Phase 2 Randomized Clinical Trial. JAMA Ophthalmol. 2018 Jan 1;136(1):29-38. doi: 10.1001/jamaophthalmol.2017.4914. PMID 29127949
- [Result] Neto HO, Regatieri CV, Nobrega MJ, Muccioli C, Casella AM, Andrade RE, Maia M, Kniggendorf V, Ferreira M, Branco AC, Belfort R Jr. Multicenter, Randomized Clinical Trial to Assess the Effectiveness of Intravitreal Injections of Bevacizumab, Triamcinolone, or Their Combination in the Treatment of Diabetic Macular Edema. Ophthalmic Surg Lasers Imaging Retina. 2017 Sep 1;48(9):734-740. doi: 10.3928/23258160-20170829-08. PMID 28902334
- [Result] Brown DM, Nguyen QD, Marcus DM, Boyer DS, Patel S, Feiner L, Schlottmann PG, Rundle AC, Zhang J, Rubio RG, Adamis AP, Ehrlich JS, Hopkins JJ; RIDE and RISE Research Group. Long-term outcomes of ranibizumab therapy for diabetic macular edema: the 36-month results from two phase III trials: RISE and RIDE. Ophthalmology. 2013 Oct;120(10):2013-22. doi: 10.1016/j.ophtha.2013.02.034. Epub 2013 May 22. PMID 23706949
- [Result] Shah AR, Yonekawa Y, Todorich B, Van Laere L, Hussain R, Woodward MA, Abbey AM, Wolfe JD. Prediction of Anti-VEGF Response in Diabetic Macular Edema After 1 Injection. J Vitreoretin Dis. 2017 May;1(3):169-174. doi: 10.1177/2474126416682569. Epub 2017 Feb 1. PMID 29104958